CLINICAL TRIAL: NCT04469595
Title: A Randomized, Masked, Controlled Study of Intravitreal ILUVIEN® Implant as Baseline Therapy in Patients With Early Diabetic Macular Edema (DME)
Brief Title: A Study of Intravitreal ILUVIEN® Implant as Baseline Therapy in Patients With Early Diabetic Macular Edema (DME)
Acronym: NEW DAY
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-20-005
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Macular Edema
Keywords: DME; CI-DME; Diabetic Macular Edema; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Fluocinolone Acetonide; Drug Implants; aflibercept

STUDY DESIGN:
Intervention Model Description: Randomized, masked, active-controlled, multi-center study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ILUVIEN Arm (Active Comparator): Intravitreal ILUVIEN
  Interventions: Drug: Iluvien 0.19 MG Drug Implant; Drug: Aflibercept
- Aflibercept Arm (Active Comparator): Intravitreal aflibercept
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Iluvien 0.19 MG Drug Implant — 0.19 mg Fluocinolone Acetonide Intravitreal Implant
  Other Names: ILUVIEN
  Arms: ILUVIEN Arm
Drug: Aflibercept — 2 mg/0.05 mL Aflibercept Anti-VEGF intravitreal injection
  Other Names: Eylea

SUMMARY:
This is a randomized, masked, active-controlled, parallel-group, multi-center study that will assess the efficacy of ILUVIEN as a baseline therapy in the treatment of Center Involving DME (CI-DME). The study will enroll patients who are either treatment naïve or have not received any DME treatments for the preceding 12 months as documented in medical records. Patients who received DME treatment >12 months before screening, must not have received >4 intravitreal injections. The study will compare 2 treatment regimens: ILUVIEN intravitreal implant (0.19 mg) followed by supplemental aflibercept as needed per protocol criteria (2 mg/0.05 mL), compared to intravitreal aflibercept loading dose (2 mg administered by intravitreal injection every 4 weeks for 5 consecutive doses) followed by supplemental aflibercept as needed per protocol criteria (2 mg/0.05 mL).

ELIGIBILITY:
Major Inclusion Criteria:

1. Male or female subjects ≥18 years of age at the time of consent.
2. Must have CI-DME confirmed by Spectral Domain Ocular Coherence Tomography (SD-OCT) and Center Subfield Thickness (CST) of: ≥350 µm in the study eye.
3. Best Corrected Visual Acuity (BCVA) of ≤80 ETDRS Letters and ≥35 ETDRS letters in the study eye at Screening Visit.

Major Exclusion Criteria:

1. Patients with Proliferative Diabetic Retinopathy (PDR); high risk proliferative diabetic retinopathy in the study eye and related complications.
2. History or current diagnosis of glaucoma or ocular hypertension (OHT) or a cup to disc ratio >0.8; History of uncontrolled intraocular pressure (defined as IOP ≥25 mmHg with maximum topical and systemic medical hypotensive treatment) or previous filtration surgery in the study eye at Screening Visit.
3. Other conditions that can cause macular edema.
4. Patients who received prior LASER photocoagulation therapy including macular grid or pan retina photocoagulation (PRP) at any time in the study eye. Prior focal LASER photocoagulation therapy outside the macula is allowed.
5. Patients who received the following therapies in the study eye:

   1. Intravitreal or periocular steroids;
   2. Intravitreal injection of aflibercept, brolucizumab, or conbercept ≤12 months prior to Screening Visit
6. Patients who received >1 intravitreal injection of ranibizumab or bevacizumab in the last 12 months; or have received ranibizumab or bevacizumab ≤6 weeks prior to Screening Visit
7. Patients who have lens opacities due to cataract or other etiologies that would make it difficult to examine the fundus or that affect the patients Activities of Daily Living (ADL).
8. Steroid Challenge Exclusion Criterion- At the Baseline Visit, patients who are determined to have an IOP ≥25 mmHg or an increase ≥8 mmHg from Screening will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The mean total number of supplemental aflibercept injections needed during the study | Baseline to 18 months
  The mean total number of supplemental aflibercept injections needed during

SECONDARY OUTCOMES:
Proportion of subjects with 15, 10 and 5 letter (ETDRS) gains from baseline | At 18 months
  Proportion of subjects with 15, 10 and 5 letter (ETDRS) gains from baseline
Area under the curve (AUC) of Best Corrected Visual Acuity (BCVA) | Baseline to 18 months
  Area under the curve (AUC) of Best Corrected Visual Acuity (BCVA)
Mean change from baseline in Center Subfield Thickness (CST) | Baseline to 18 months
  Mean change from baseline in Center Subfield Thickness (CST)
Area under the curve (AUC) of Center Subfield Thickness (CST) | Baseline to 18 months
  Area under the curve (AUC) of Center Subfield Thickness (CST)
Mean change from baseline in the National Eye Institute Visual Function Questionnaire (NEI VFQ-25) composite score and subscale scores | At 18 months
  The NEI VFQ-25 is a questionnaire that allows the individual to report on their level of visual function. Scores range from 0-100, with a score of 0 being the worst outcome and 100 being the best outcome.
Safety Outcome Endpoints: The incidence and severity of treatment-related adverse events | Baseline to 18 months
  The incidence and severity of treatment-related adverse events

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Investigative Site, Phoenix, Arizona
  - Investigative Site, Tucson, Arizona
  - Investigative Site, Beverly Hills, California
  - Investigative Site, Glendale, California
  - Investigative Site, Laguna Hills, California
  - Investigative Site, Santa Ana, California
  - Investigative Site, Colorado Springs, Colorado
  - Investigative Site, Clearwater, Florida
  - Investigative Site, Orlando, Florida
  - Investigative Site, Palm Beach Gardens, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, Marietta, Georgia
  - Investigative Site, Sandy Springs, Georgia
  - Investigative Site, Elmhurst, Illinois
  - Investigative Site, Lemont, Illinois
  - Investigative Site, Oak Park, Illinois
  - Investigative Site, Springfield, Illinois
  - Investigative Site, Leawood, Kansas
  - Investigative Site, Shawnee Mission, Kansas
  - Investigative Site, West Monroe, Louisiana
  - Investigative Site, Baltimore, Maryland
  - Investigative Site, Detroit, Michigan
  - Investigative Site, Grand Blanc, Michigan
  - Investigative Site, Independence, Missouri
  - Investigative Site, Bloomfield, New Jersey
  - Investigative Site, Beachwood, Ohio
  - Investigative Site, Cincinnati, Ohio
  - Investigative Site, Cleveland, Ohio
  - Investigative Site, Youngstown, Ohio
  - Investigative Site, Tulsa, Oklahoma
  - Investigative Site, Erie, Pennsylvania
  - Investigative Site, Columbia, South Carolina
  - Investigative Site, Dallas, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, McAllen, Texas
  - Investigative Site, San Antonio, Texas
  - Investigative Site, The Woodlands, Texas
  - Investigative Site, Roanoke, Virginia
  - Investigative Site, Warrenton, Virginia

IPD SHARING:
Plan to Share IPD: No